CLINICAL TRIAL: NCT05422508
Title: A Double-blind, Randomized, Multi-Center, Active Controlled Phase 2 Clinical Trial to Evaluate the Safety and Immunogenicity After MG1111(BARICELA Inj.) as 2nd Vaccination in 4 ~ 6 Year Old Healthy Children With a History of 1st Varicella Vaccination
Brief Title: Evaluate the Safety and Immunogenicity After MG1111(BARICELA Inj.) as 2nd Vaccination in 4 ~ 6 Year Old Healthy Children With a History of 1st Varicella Vaccination
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: MG1111_VAR_P0201
Record Dates: First submitted 2022-05-24; First posted 2022-06-16 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Varicella
MeSH Terms: conditions — Chickenpox | interventions — Chickenpox Vaccine

STUDY DESIGN:
Intervention Model Description: After the Protocol v4.1 was approved by Ministry of Food and Drug Safety (02Jun2023), Subject eligibility was change to 4 ~ 6 Year Old Healthy Children With a History of 1st Varicella Vaccination instead of 1st SUDUVAX inj. and Active Comparator: VARIVAX arm was deleted.
  *VARIVAX release has been discontinued.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MG1111(BARICELA) arm (Experimental): 0.5ml, single dose, subcutaneous injection
  Interventions: Biological: MG1111 (BARICELA)
- VARIVAX arm (Active Comparator): 0.5ml, single dose, subcutaneous injection
  Interventions: Biological: VARIVAX
- Suduvax arm (Active Comparator): 0.5ml, single dose, subcutaneous injection
  Interventions: Biological: Suduvax

INTERVENTIONS:
Biological: MG1111 (BARICELA) — 0.5ml, single dose, subcutaneous injection
  Arms: MG1111(BARICELA) arm
Biological: VARIVAX — 0.5ml, single dose, subcutaneous injection
  Arms: VARIVAX arm
Biological: Suduvax — 0.5ml, single dose, subcutaneous injection
  Arms: Suduvax arm

SUMMARY:
* Primary objective is to assess the safety of MG1111 until Day 42 using as 2nd vaccination
* Secondary objective to assess the immunogenicity and safety of MG1111 using as 2nd vaccination

DETAILED DESCRIPTION:
1. Safety

   * Incidence of fever (temperature ≥39.0℃) within 42 days after the IP administration
   * Incidence of fever (temperature ≥39.0℃) within 7 days after the IP administration
   * Solicited local/systemic AEs occurred within 7 days after the IP administration
   * Unsolicited adverse events that occurred within 42 days after the IP administration
   * Serious adverse events that occurred within 1 year after the IP administration
   * Vital signs and physical examinations
2. Efficacy (Immunogenicity)

   -GMT(Geometric Mean Titer) and GMR(Geometric Mean Ratio(fold change))measured by the glycoprotein enzyme-linked immunosorbent assay (gpELISA) at before and 42 days after the IP administration
3. Exploratory assessment

   * GMV and GMR of VZV-CMI response measured by INF-r ELISPOT at before and 42 days after the IP administration
   * GMT and GMR of the antibody titer measured by gpELISA at before and after the IP administration for 3 years
   * Varicella-like rash and Varicella-zoster virus genotyping analysis occurred after IP administration for 3 years

ELIGIBILITY:
Inclusion Criteria:

* Healthy children between 4 and 6 years of age as of the date of written consent
* Subjects who have a history of 1st Varicella vaccination at least 3 years ago from the administration of investigational product
* Subjects or parent/legal representative willing to provide written informed consent and able to comply with the study requirements
* Negative history of Varicella infection

Exclusion Criteria:

* Subjects with a history of exposure to varicella through contact with a varicella patient at home, school, or childcare facility within 4 weeks before the administration of investigational drug
* Subjects who have a history 2 times or more of varicella vaccine injections
* Subjects who had an acute febrile (at least 38.0 ℃) episode at some time during the 72 hours before the administration of investigational product
* Subjects who had any suspected allergy symptoms including systemic rash during the 72 hours before the administration of investigational product
* Subjects with a history of Guillain-Barre syndrome.
* Subjects with a severe chronic disease and considered ineligible for the study at Investigator's discretion
* Subjects with a history of hypersensitivity to any ingredient such as gelatin, antibiotics (Neomycin, Kanamycin, Erythromycin)
* Active tuberculosis patient
* Subjects who had received other vaccinations within 4 weeks before the administration of investigational product
* Subjects with immunodeficiency history
* Subjects who had received salicylates (aspirin, bismuth, subsalicylates) within 4 weeks before the administration of investigational drug
* Subjects who administered immune globulin, gamma globulin, or blood products such as whole blood within 44 weeks before the administration of investigational drug
* Subjects who had received immunosuppressant or immune modifying drug within 12 weeks before the administration of investigational drug
* A. Azathioprine, Cyclosporin, Interferon, G-CSF, Tacrolimus, Everolimus, Sirolimus, etc.
* B. Subjects who administered high dose of corticosteroids (greater than 2 mg/kg/day in case of under 10kg subjects or ≥20mg/day in case of above 10kg subject of prednisone for 14 days) (However, inhaled, intranasal, topical corticosteroids administration in allowed)
* Subjects who administered anti-viral drug within 4 weeks before the administration of investigational drug
* Subjects who have participated in any other clinical trials within 24 weeks of the administration of the investigational product
* Subjects with other clinically significant medical or psychological condition who are considered by the Investigator to be ineligible for the study

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 230 (Estimated)
Dates: Start 2022-07-05 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of fever (temperature ≥39.0℃) | within 7 days
  Incidence of fever (temperature ≥39.0℃) within 7days after the IP administration
Solicited local / systemic adverse events | within 7 days
  Solicited local / systemic adverse events that occurred within 7 days after the IP administration
Unsolicited adverse events | within 42 days
  Unsolicited adverse events that occurred within 42 days after the IP administration
Vital signs (blood pressure, pulse rate, respiration rate and body temperature) | within 42 days
  descriptive statistics (number of subjects, mean, standard deviation, median, minimum, and maximum) of change from baseline to 42 days will be presented for each group.
Incidence of fever (temperature ≥39.0℃) | within 42days
  Incidence of fever (temperature ≥39.0℃) within 42 days after the IP administration
Physical examinations (Cardiovascular, respiratory, gastrointestinal, liver, metabolic/endocrine, kidney, reproductive, musculoskeletal and nervous system, head/neck, and skin) | within 42 days
  the change from baseline to 42 days will be classified into 'normal/abnormal, not clinically significant (NCS)' or 'abnormal, clinically significant (CS)', and the frequency and percentage are presented in a shift table.

SECONDARY OUTCOMES:
Serious adverse events | within 1 year
  Serious adverse events that occurred within 1 year after the IP administration
GMT and GMR of the antibody titer | at Day1, Day42
  GMT and GMR of the antibody titer measured by gpELISA at before and 42 days after the IP administration

OTHER OUTCOMES:
GMV and GMR of VZV-CMI response | at Day1, Day42
  GMV and GMR of VZV-CMI response measured by INF-r ELISPOT at before and 42 days after the IP administration
GMT and GMR of the antibody titer | at Year1, Year2, Year3
  GMT and GMR of the antibody titer measured by gpELISA at before and after the IP administration for 3 year
Varicella-like rash | anytime within 3 years (if applicable)
  Varicella-like rash occurred after IP administration for 3 years
Varicella-zoster virus genotyping | anytime within 3 years (if applicable)
  Varicella-zoster virus genotyping analysis occurred after IP administration for 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Yun-kyung Kim, M.D., Ph.D, Principal Investigator — Korea University Ansan Hospital
Locations (1):
- Korea University Ansan Hospital, Ansan, South Korea